CLINICAL TRIAL: NCT06294665
Title: Comparison Between Bupivacaine-Dexmedetomidine Versus Bupivacaine-Dexamethasone in Pericapsular Nerve Group (PENG) Block as Post-operative Analgesia in Hip Surgeries.
Brief Title: Comparison Between Bupivacaine-Dexmedetomidine Versus Bupivacaine-Dexamethasone in Pericapsular Nerve Group (PENG) Block
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD113/2023
Record Dates: First submitted 2024-02-28; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Hip Fractures; Post Operative Pain
MeSH Terms: conditions — Hip Fractures; Pain, Postoperative | interventions — Dental Occlusion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A : ( Bupivacaine + Dexmedetomidine ) (Active Comparator): Group A : will receive bupivacaine 0.25% + dexmedetomidine 1 mic/kg, total volume (20 ml)
  Interventions: Drug: Pericapsular Nerve Group (PENG) Block
- Group B: ( Bupivacaine + Dexamethasone ) (Active Comparator): Group B : will receive bupivacaine 0.25% +dexamethasone (8 mg), total volume(20 ml).
  Interventions: Drug: Pericapsular Nerve Group (PENG) Block

INTERVENTIONS:
Drug: Pericapsular Nerve Group (PENG) Block — The PENG block will be performed ,the patient is placed in the supine position , the procedural leg is slightly abducted, the curvilinear low-frequency ultrasound probe will be placed over the line parallel to the inguinal ligament. It will subsequently rotated 45◦ to identify the anterior inferior iliac spine, the iliopubic eminence, and the psoas tendon. A 22-gauge, 80 mm echogenic needle will inserted in an in-plane approach to place the tip in the musculofascial plane between the pubic ramus posteriorly and the psoas tendon anteriorly. Following negative aspiration, by one of the two syringes each one has a serial number corresponding to each group.

SUMMARY:
The aim of this work is to compare the effectiveness of bupivacaine- dexmedetomidine mixture versus bupivacaine-dexamethasone mixture in PENG Block as Post-operative Analgesia in Hip surgeries

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years.
2. Sex: Both sexes.
3. American Society of Anaesthesiologists (ASA) Physical Status Class I and II.
4. Scheduled for hip surgeries under spinal anaesthesia.

Exclusion Criteria:

1. Declining to give written informed consent.
2. History of allergy to the medications used in the study.
3. Contraindications to regional anesthesia (including patient refusal, coagulopathy and local infection).
4. Psychiatric disorder.
5. American Society of Anesthesiologists (ASA) Physical Status Class III and IV.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
The time to the first request of analgesia | 9 months
  The time interval between the onset of the local infiltration done at the end of the operation and the first request to postoperative analgesia.

SECONDARY OUTCOMES:
Total doses of analgesia (Nalbuphine) given to patients in 24 hours postoperatively | 9 months
Occurrence of side effects of drugs. | 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt